CLINICAL TRIAL: NCT03087955
Title: Efficacy and Safety Study of Acoziborole (SCYX-7158) in Patients With Human African Trypanosomiasis (HAT) Due to Trypanosoma Brucei Gambiense: a Multicentre, Open-label, Prospective Study
Brief Title: Efficacy and Safety of Acoziborole (SCYX-7158) in Patients With Human African Trypanosomiasis Due to T.b. Gambiense
Acronym: OXA002
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNDi-OXA-02-HAT
Record Dates: First submitted 2017-03-07; First posted 2017-03-23 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Trypanosomiasis, African; Gambiense Trypanosomiasis; Sleeping Sickness
MeSH Terms: conditions — Trypanosomiasis, African | interventions — SCYX 7158

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Late-stage HAT (Experimental): Participants with confirmation of HAT by detection of the parasite in the blood and/or lymph and/or cerebrospinal fluid (CSF) at the investigational center. If testing for parasites in CSF was negative, the CSF white blood cell count, measured at the investigational center, had to be above 20 cells/µL for classification as late-stage HAT. Participants received 960 mg acoziborole as a single oral dose.
  Interventions: Drug: Acoziborole
- Early- and intermediate-stage HAT (Experimental): Participants with confirmation of HAT by detection of the parasite in the blood and/or lymph at the investigational center. Parasites had to be absent from the CSF. The CSF white blood cell count, measured at the investigational center, had to be between 6 and 20 cells/µL for classification as intermediate stage HAT and equal to or below 5 cells/µL for classification as early-stage HAT. Participants received 960 mg acoziborole as a single oral dose.
  Interventions: Drug: Acoziborole

INTERVENTIONS:
Drug: Acoziborole — Acoziborole 3 x 320 mg tablets (fasted state)
  Other Names: SCYX-7158

SUMMARY:
The goal of this study is to assess efficacy and safety of acoziborole in adult participants with Trypanosoma brucei gambiense (T.b. gambiense) HAT, either early- or intermediate-stage HAT (first arm) or late-stage HAT (second arm). Participants will receive 3 tablets of 320 mg as a single oral dose of acoziborole in the fasting state on Day 1. Participants will stay in the hospital for observation for 15 days. In total, participants will be followed for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient
* 15 years of age or older
* Signed informed consent form (as well as assent from illiterate and under-age patients, and those unable to give consent)
* Karnofsky Performance Status above 50
* Able to ingest oral tablets
* Having a permanent address or being traceable by other persons
* Able to comply with the schedule of follow-up visits and requirements of the study
* Agreement to be hospitalised in order to receive treatment
* For patients with late-stage HAT:

  * Confirmation of g-HAT by detection of the parasite in the blood and/or the lymph and/or the CSF, at the investigational centre
  * If trypanosomes are found in the blood or lymph, but not in the CSF, the CSF WBC, measured at the investigational centre, must be above 20/μL for the patient to be included in the cohort of patients with late-stage HAT
* For patients with early- or intermediate-stage HAT:

  * Confirmation of g-HAT by detection of the parasite in the blood and/or the lymph, at the investigational centre
  * Absence of parasites in the CSF
  * The CSF WBC, measured at the investigational centre, must be between 6 and 20/μL for the patient to be included in the cohort of patients with intermediate-stage HAT and equal to or below 5/μL for the patient to be included in the cohort of patients with early-stage HAT.

Exclusion Criteria:

* Severe malnourishment, defined as body-mass index (BMI) below 16
* Pregnancy or breastfeeding (for women of child-bearing potential, confirmed pregnancy on a urine pregnancy test performed within 24 hours prior to administration of acoziborole)
* Clinically significant medical condition that could, in the opinion of the Investigator, jeopardise the patient's safety or interfere with participation in the study, including, but not limited to significant liver or cardiovascular disease, suspected or proven active infection, central nervous system trauma or seizure disorder, coma or consciousness disturbances
* Severely deteriorated health status, e.g. due to cardiovascular shock, respiratory distress syndrome or end-stage disease
* Previously treated for HAT (except prior treatment with pentamidine)
* Prior enrolment in the study
* Foreseeable difficulty complying with follow-up, including migrant worker, refugee status, itinerant trader etc.
* Current alcohol abuse or drug addiction
* Not tested for malaria and/or not having received appropriate treatment for malaria
* Not having received appropriate treatment for soil-transmitted helminthiasis
* Clinically significant abnormal laboratory values including aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) more than 2 times the upper limit of normal (ULN), total bilirubin more than 1.5 ULN, severe leukopenia at less than 2000/mm^3, Potassium below 3.5 mmol/L, any other clinically significant abnormal laboratory value

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Kande Betu Kumeso, Dr, Principal Investigator — Ministère de la Santé, The Democratic Republic of the Congo
Locations (12):
- Democratic Republic of the Congo (11):
  - Centre de Traitement de Nkara, Nkara, Bandundu
  - Centre de Traitement de Kimpese, Kimpese, Bas-Congo Province
  - Hôpital Général de Référence de Ngandajika, Gandajika, East Kasai
  - Hôpital Secondaire de Katanda, Katanda, East Kasai
  - Hôpital de Dipumba, Mbuji-Mayi, East Kasai
  - Hôpital Général de Référence de Bagata, Bagata, Kwilu
  - Hôpital Général de Référence de Masi-Manimba, Masi-Manimba, Kwilu
  - Hôpital Général de Référence de Kwamouth, Kwamouth, Mai Ndombe
  - Hopital Général de Réference de Bandundu, Bandundu Province
  - Hôpital de Référence d'Isangi, Isangi
  - Hôpital Général de Référence Roi Baudouin, Kinshasa
- Centre de Traitement de la THA de Dubreka, Dubréka, Dubreka, Guinea

IPD SHARING:
Plan to Share IPD: Yes
The data underlying the results of this study are available upon request because they contain potentially sensitive personal information, which must be de-identified at the individual level. Interested researchers may request access to de-identified participant data from Vivli, the data-sharing partner of the DNDi, commissioner of this study, at https://vivli.org/ourmember/dndi/.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Available upon request (see above)
Access Criteria: Available upon request (see above)
URL: https://vivli.org/ourmember/dndi/

REFERENCES:
- [Result] Betu Kumeso VK, Kalonji WM, Rembry S, Valverde Mordt O, Ngolo Tete D, Pretre A, Delhomme S, Ilunga Wa Kyhi M, Camara M, Catusse J, Schneitter S, Nusbaumer M, Mwamba Miaka E, Mahenzi Mbembo H, Makaya Mayawula J, Layba Camara M, Akwaso Massa F, Kaninda Badibabi L, Kasongo Bonama A, Kavunga Lukula P, Mutanda Kalonji S, Mariero Philemon P, Mokilifi Nganyonyi R, Embana Mankiara H, Asuka Akongo Nguba A, Kobo Muanza V, Mulenge Nasandhel E, Fifi Nzeza Bambuwu A, Scherrer B, Strub-Wourgaft N, Tarral A. Efficacy and safety of acoziborole in patients with human African trypanosomiasis caused by Trypanosoma brucei gambiense: a multicentre, open-label, single-arm, phase 2/3 trial. Lancet Infect Dis. 2023 Apr;23(4):463-470. doi: 10.1016/S1473-3099(22)00660-0. Epub 2022 Nov 29. PMID 36460027

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at Human African Trypanosomiasis (HAT) treatment centers in the Democratic Republic of Congo and Guinea. A total of 260 HAT-positive participants signed informed consent and 208 participants (167 with late- and 41 with early- and intermediate-stage HAT) were included in the study and treated. 52 participants were not included, mainly due to exclusion criteria met and/or inclusion criteria not met. Participants were enrolled between 11 October 2016 and 25 March 2019.
Pre-assignment Details: The pre-treatment period of up to 15 days included pre-screening, screening, and treatment of concurrent malaria/soil-transmitted helminthiasis. At the end of this period, all participants (regardless of HAT-stage) were treated with acoziborole.
Groups:
- Late-stage HAT: Participants with confirmation of HAT by detection of the parasite in the blood and/or lymph and/or cerebrospinal fluid (CSF) at the investigational center. If testing for parasites in CSF was negative, the CSF white blood cell count, measured at the investigational center, had to be above 20 cells/µL for classification as late-stage HAT. Participants received 960 mg acoziborole as a single oral dose.
  Acoziborole: Acoziborole 960 mg as a single oral dose (3 x 320 mg tablets; fasted state)
- Early- and Intermediate-stage HAT: Participants with confirmation of HAT by detection of the parasite in the blood and/or lymph at the investigational center. Parasites had to be absent from the CSF. The CSF white blood cell count, measured at the investigational center, had to be between 6 and 20 cells/µL for classification as intermediate stage HAT and equal to or below 5 cells/µL for classification as early-stage HAT. Participants received 960 mg acoziborole as a single oral dose.
  Acoziborole: Acoziborole 960 mg as a single oral dose (3 x 320 mg tablets; fasted state)
Period: Overall Study
Arm/Group | Late-stage HAT | Early- and Intermediate-stage HAT
Started | 167 | 41
Completed | 160 | 41
Not Completed | 7 | 0
Not completed — Death | 4 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Late-stage HAT | Early- and Intermediate-stage HAT | Total
Number analyzed (Participants) | 167 | 41 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (11.2) | 40.9 (15.0) | 34.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 26 | 91
  Male | 102 | 15 | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Sub-Saharan African | 167 | 41 | 208
Region of Enrollment [Number; unit: participants]
  Guinea | 27 | 7 | 34
  Congo, The Democratic Republic of the | 140 | 34 | 174
White blood cells (WBC) in cerebrospinal fluid (CSF) [Mean (Standard Deviation); unit: cells/µL] | 398.8 (438.4) | 7.8 (5.3) | 321.3 (422.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Late-stage HAT Whose Treatment Outcome Was a Success at Month 18 According to Adapted World Health Organization (WHO) Criteria
Description: Success was defined according to an algorithm based on the criteria adapted from the WHO Recommendations of the Informal Consultation on Issues for Clinical Product Development for Human African Trypanosomiasis 2007 (WHO/CDS/NTD/IDM/2007.1). Success was defined as a cure or a probable cure. Failure was defined as a relapse, probable relapse, death, use of rescue medication, loss to follow-up, refusal of all post-treatment lumbar puncture, and, in the absence of lumbar puncture at the Month 18 visit, an unfavorable outcome earlier than Month 18, or signs and symptoms evoking a relapse at Month 18. An estimate of the percentage of participants whose treatment outcome was a success at Month 18 and the 95% Jeffreys confidence interval (CI) of the estimate were provided.
Time Frame: 18 months post-dose
Population: The modified intention-to-treat (mITT) set included all participants who received at least 1 tablet of acoziborole, excluding participants who fled the region due to armed conflict or natural disaster or due to force majeure and for whom no failure was detected early* and no data were available at Month 12 and Month 18.** * Parasite, need for rescue medication, death, or more than 50 WBC/μL in CSF at Month 6.
  ** Due to armed conflict, natural disaster, or force majeure affecting the site.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Late-stage HAT
Number analyzed (Participants) | 167
percentage of participants | 95.2 [91.2 to 97.7]

2. Secondary Outcome: Percentage of Participants With Late-stage HAT Whose Treatment Outcome Was a Success at Month 12 According to Adapted WHO Criteria
Description: Success was defined according to an algorithm based on the criteria adapted from the WHO Recommendations of the Informal Consultation on Issues for Clinical Product Development for Human African Trypanosomiasis 2007 (WHO/CDS/NTD/IDM/2007.1). Success was defined as a cure or a probable cure. Failure was defined as a relapse, probable relapse, death, use of rescue medication, loss to follow-up, refusal of all post-treatment lumbar puncture, and, in the absence of lumbar puncture at the end of Month 12, an unfavorable outcome earlier than end of Month 12, or signs and symptoms evoking a relapse at end of Month 12. For participants who continued after Month 12, data after Month 12 were considered in the algorithm. An estimate of the percentage of participants whose treatment outcome was a success at Month 12 and the 95% Jeffreys CI of the estimate were provided.
Time Frame: 12 months post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Late-stage HAT
Number analyzed (Participants) | 167
percentage of participants | 95.8 [91.9 to 98.1]

3. Secondary Outcome: Percentage of Participants With Late-stage HAT Whose Treatment Outcome Was a Success at Month 6 According to Adapted WHO Criteria
Description: Success was defined according to an algorithm based on to the criteria adapted from the WHO Recommendations of the Informal Consultation on Issues for Clinical Product Development for Human African Trypanosomiasis 2007 (WHO/CDS/NTD/IDM/2007.1). Success was defined as a cure or a probable cure. Failure was defined as a relapse, probable relapse, death, use of rescue medication, loss to follow-up, refusal of all post-treatment lumbar puncture, and, in the absence of lumbar puncture at the end of Month 6, an unfavorable outcome earlier than end of Month 6, or signs and symptoms evoking a relapse at end of Month 6. For participants who continued after Month 6, data after Month 6 were considered in the algorithm. An estimate of the percentage of participants whose treatment outcome was a success at Month 6 and the 95% Jeffreys CI of the estimate were provided.
Time Frame: 6 months post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Late-stage HAT
Number analyzed (Participants) | 167
percentage of participants | 94.6 [90.4 to 97.3]

4. Secondary Outcome: Percentage of Participants With Early- and Intermediate-stage HAT Whose Treatment Outcome Was a Success at Month 18 According to Adapted WHO Criteria
Description: Success was defined according to an algorithm based on the criteria adapted from the WHO Recommendations of the Informal Consultation on Issues for Clinical Product Development for Human African Trypanosomiasis 2007 (WHO/CDS/NTD/IDM/2007.1). Success was defined as a cure or a probable cure. Failure was defined as a relapse, probable relapse, death, use of rescue medication, loss to follow-up, refusal of all post-treatment lumbar puncture, and, in the absence of lumbar puncture at the end of Month 18, an unfavorable outcome earlier than end of Month 18, or signs and symptoms evoking a relapse at end of Month 18. An estimate of the percentage of participants whose treatment outcome was a success at Month 18 and the 95% Jeffreys CI of the estimate were provided.
Time Frame: 18 months post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Early- and Intermediate-stage HAT
Number analyzed (Participants) | 41
percentage of participants | 100.0 [94.1 to 100.0]

5. Secondary Outcome: Percentage of Participants With Early- and Intermediate-stage HAT Whose Treatment Outcome Was a Success at Month 12 According to Adapted WHO Criteria
Description: as for outcome 2
Time Frame: 12 months post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Early- and Intermediate-stage HAT
Number analyzed (Participants) | 41
percentage of participants | 100.0 [94.1 to 100.0]

6. Secondary Outcome: Percentage of Participants With Early- and Intermediate-stage HAT Whose Treatment Outcome Was a Success at Month 6 According to Adapted WHO Criteria
Description: Success was defined according to an algorithm based on the criteria adapted from the WHO Recommendations of the Informal Consultation on Issues for Clinical Product Development for Human African Trypanosomiasis 2007 (WHO/CDS/NTD/IDM/2007.1). Success was defined as a cure or a probable cure. Failure was defined as a relapse, probable relapse, death, use of rescue medication, loss to follow-up, refusal of all post-treatment lumbar puncture, and, in the absence of lumbar puncture at the end of Month 6, an unfavorable outcome earlier than end of Month 6, or signs and symptoms evoking a relapse at end of Month 6. For participants who continued after Month 6, data after Month 6 were considered in the algorithm. An estimate of the percentage of participants whose treatment outcome was a success at Month 6 and the 95% Jeffreys CI of the estimate were provided.
Time Frame: 6 months post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Early- and Intermediate-stage HAT
Number analyzed (Participants) | 41
percentage of participants | 100.0 [94.1 to 100.0]

7. Secondary Outcome: Estimated Percentage of Participants With Late-stage HAT Whose Treatment Outcome Was Not a Proven Failure at Month 18, Based on the Kaplan-Meier Analysis of Time to Proven and Definitive Failure
Description: Failure was defined as the first objective evidence of proven and definitive (sustainable) failure, defined as death; rescue medication use; trypanosomes in any body fluid at Month 6, 12, or 18; a cerebrospinal fluid (CSF) white blood cell count (WBC) of >50 cells/μL at Month 6 followed by confirmation of failure (defined as CSF WBC >20 cells/μL at Month 12 and/or Month 18 and/or signs and symptoms evoking a relapse at Month 12 and/or Month 18); a CSF WBC >20 cells/μL at Month 12 followed by confirmation of failure (defined as CSF WBC >20 cells/μL at Month 18 and/or signs and symptoms evoking a relapse at Month 18); or a CSF WBC >20 cells/μL at Month 18. This outcome was analyzed using a Kaplan-Meier approach to estimate the cumulative rate of proven and definitive failures. The proven failure-free probability was estimated as an alternative (more liberal) success rate (95% CI) at Month 18 based on the Kaplan-Meier estimate of the rate of participants who were not proven failures
Time Frame: 18 months post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Late-stage HAT
Number analyzed (Participants) | 167
percentage of participants | 96.0 [91.0 to 98.0]

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Occurrence of any AEs, during the observation period and until 6 months post-dose (for non-serious AEs) and until 18 months post-dose for SAEs. Analysis of AEs was based on the concept of TEAEs, defined as any AEs occurring on or after the date of study-drug administration or worsening in intensity on or after the date of study-drug administration.
Time Frame: From the single dose acoziborole administration until 6 months post-dose for non-serious AEs and 18 months post-dose for serious AEs
Population: The Treated set included all participants who received at least one tablet of acoziborole.
Measure: Count of Participants; unit: Participants
Groups:
- Late-stage HAT: Participants with confirmation of HAT by detection of the parasite in the blood and/or lymph and/or cerebrospinal fluid (CSF) at the investigational center. If testing for parasites in CSF was negative, the CSF white blood cell count, measured at the investigational center, had to be above 20 cells/μL for classification as late-stage HAT. Participants received 960 mg acoziborole as a single oral dose.
  Acoziborole: Acoziborole 960 mg as a single oral dose (3 x 320 mg tablets; fasted state)
- Early- and Intermediate-stage HAT: Participants with confirmation of HAT by detection of the parasite in the blood and/or lymph at the investigational center. Parasites had to be absent from the CSF. The CSF white blood cell count, measured at the investigational center, had to be between 6 and 20 cells/μL for classification as intermediate stage HAT and equal to or below 5 cells/μL for classification as early-stage HAT. Participants received 960 mg acoziborole as a single oral dose.
  Acoziborole: Acoziborole 960 mg as a single oral dose (3 x 320 mg tablets; fasted state)
- Any Stage HAT: Participants with any stage HAT, including all participants irrespective of HAT stage (participants with late-stage HAT and participants with early- and intermediate-stage HAT). Participants received 960 mg acoziborole as a single oral dose.
Arm/Group | Late-stage HAT | Early- and Intermediate-stage HAT | Any Stage HAT
Number analyzed (Participants) | 167 | 41 | 208
Participants | 127 | 28 | 155

9. Secondary Outcome: Number of Participants With Serious TEAEs
Description: Occurrence of any serious TEAEs during the observation period and until 18 months post-dose.
Time Frame: From the single dose acoziborole administration until 18 months post-dose
Population: The Treated set included all participants who received at least one tablet of acoziborole.
Measure: Count of Participants; unit: Participants
Arm/Group | Late-stage HAT | Early- and Intermediate-stage HAT | Any Stage HAT
Number analyzed (Participants) | 167 | 41 | 208
Participants | 18 | 3 | 21

10. Secondary Outcome: Acoziborole Area Under the Curve From Time Zero to 240 Hours Post Dose (AUC0-240h) in Whole Blood Considering Concentration-time Data up to 240 Hours After a Single Administration
Description: Participants received a single dose of 960 mg acoziborole on Day 1. Acoziborole in whole blood was assessed pre-dose and 4, 9, 24, 48, 72, 96, and 240 hours after the single administration, (on Days 1, 2, 3, 4, 5, and 11). Data up to 240 hours post dose were considered for this analysis. Descriptive statistics of the AUC0-240h were presented. The activity of acoziborole is more exposure-dependent than concentration-dependent, therefore the exposure (AUC) was used as the main PK data for efficacy purposes.
Time Frame: Pre-dose and 4, 9, 24, 48, 72, 96, and 240 hours post-dose
Population: The pharmacokinetic (PK) analysis set included participants who received an oral dose of 960 mg acoziborole, as far as the information about time and amount was available, and for whom at least one blood sample for PK was available.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Late-stage HAT | Early- and Intermediate-stage HAT | Any Stage HAT
Number analyzed (Participants) | 167 | 41 | 208
h*ng/mL | 2217617.78 (647696.87) | 2051104.88 (485620.67) | 2184795.53 (621610.31)

11. Secondary Outcome: Mean Acoziborole Concentration in CSF After 240 Hours in Participants With Late-stage HAT
Description: Participants received a single dose of 960 mg acoziborole on Day 1. Acoziborole in CSF of participants with late-stage HAT was assessed 240 hours after the single administration (on Day 11). Descriptive statistics of the acoziborole concentration were presented.
Time Frame: 240 hours post-dose
Population: The PK analysis set included participants who received an oral dose of 960 mg acoziborole, as far as the information about time and amount was available, and for whom at least one blood sample for PK was available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Late-stage HAT
Number analyzed (Participants) | 129
ng/mL | 100.8 (63.968)

12. Secondary Outcome: Mean Acoziborole Concentration in CSF After 240 Hours in Participants With Early- and Intermediate-stage HAT
Description: Participants received a single dose of 960 mg acoziborole on Day 1. Acoziborole in CSF of participants with early- and intermediate-stage HAT was assessed 240 hours after the single administration (on Day 11). Descriptive statistics of the acoziborole concentration were presented.
Time Frame: 240 hours post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Early- and Intermediate-stage HAT
Number analyzed (Participants) | 31
ng/mL | 81.4 (48.5)

ADVERSE EVENTS:
Time Frame: Non-serious AEs were recorded from the time of administration of acoziborole on Day 1 until the 6 month follow-up visit. Serious AEs were collected from the time of providing written informed consent until the end of the follow-up (Month 18). TEAEs were defined as any AEs occurring on or after the date of study-drug administration or worsening in intensity on or after the date of study-drug administration.
Description: The Investigator collected all AEs observed directly and those reported spontaneously. AEs and serious AEs were defined according to standard definitions. In specific, in this study, alanine aminotransferase or aspartic aminotransferase levels 3 times above the upper limit of normal (ULN) accompanied by total bilirubin levels 2 times above the ULN were considered serious AEs. Furthermore, any suspected transmission of an infectious agent via a medicinal product was also considered a serious AE.
Arm/Group | Late-stage HAT | Early- and Intermediate-stage HAT
All-Cause Mortality (participants affected / at risk) | 4/167 | 0/41
Serious Adverse Events (participants affected / at risk) | 18/167 | 3/41
Other Adverse Events (participants affected / at risk) | 127/167 | 27/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Late-stage HAT (N=167) | Early- and Intermediate-stage HAT (N=41)
Malaria (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Extrapulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (2) | 0 (0)
Puerperal infection (Infections and infestations) | 0 (0) | 1 (1)
Systemic infection (Infections and infestations) | 1 (1) | 0 (0)
Typhoid fever (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Brief psychotic disorder with marked stressors (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Organic brain syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Late-stage HAT (N=167) | Early- and Intermediate-stage HAT (N=41)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 4 (4) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (9) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 13 (14) | 0 (0)
Asthenia (General disorders) | 13 (14) | 5 (5)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Feeling hot (General disorders) | 2 (2) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 27 (30) | 4 (4)
Abscess (Infections and infestations) | 3 (3) | 0 (0)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 3 (3) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 5 (6) | 2 (2)
Dysentery (Infections and infestations) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 2 (2) | 0 (0)
Filariasis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (5) | 0 (0)
Helminthic infection (Infections and infestations) | 1 (1) | 1 (1)
Infection parasitic (Infections and infestations) | 3 (3) | 0 (0)
Infectious colitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 1 (1)
Malaria (Infections and infestations) | 22 (27) | 5 (5)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Schistosomiasis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Syphilis (Infections and infestations) | 2 (2) | 0 (0)
Typhoid fever (Infections and infestations) | 4 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (10) | 1 (1)
Varicella (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 5 (5) | 0 (0)
Wound infection (Infections and infestations) | 3 (3) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 21 (22) | 11 (13)
Procedural pain (Injury, poisoning and procedural complications) | 39 (46) | 13 (17)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 1 (1)
Blood sodium decreased (Investigations) | 2 (2) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 6 (6) | 0 (0)
Weight increased (Investigations) | 19 (19) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Overweight (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 1 (1)
Formication (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 39 (49) | 12 (14)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 6 (7) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 6 (6) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Bulimia nervosa (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Eating disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Enuresis (Psychiatric disorders) | 2 (5) | 0 (0)
Insomnia (Psychiatric disorders) | 13 (16) | 2 (2)
Psychotic disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The principal limitation of this study was the lack of comparator or control group, instead comparisons were made with a yardstick based on historical data. The sample size was based on the maximum feasible enrolment within a reasonable timeframe, because of the challenges of enrolling patients with HAT in clinical trials given the drastic decline in prevalence, and in order to expose as many participants to the test drug as possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor authorizes publications by a single site provided that multicentric results are published beforehand and any communication is submitted to the sponsor for review at least 28 days before the expected publication date. The sponsor can comment for 28 days. Upon sponsor request, any confidential information will have to be removed before publishing. Publishing can be postponed by 90 additional days, should the sponsor want to protect data through a patent application or any other mean.

DOCUMENTS (2):
  • Study Protocol (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT03087955/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT03087955/SAP_001.pdf